CLINICAL TRIAL: NCT03634137
Title: A Phase Ib Study to Confirm the Pharmacokinetics and Melanogenic Potential of Controlled-Release Bioresorbable Implants of Afamelanotide in Healthy Volunteers
Brief Title: Implant Pharmacokinetic and Pharmacodynamic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clinuvel Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CUV028
Record Dates: First submitted 2010-03-29; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: Afamelanotide; Nontherapeutic Human Experimentation in healthy volunteers
MeSH Terms: interventions — afamelanotide

STUDY DESIGN:
Intervention Model Description: Participants were assigned to receive either a 16 mg bioresorbable afamelanotide implant from the previous manufacturing process or a 16 mg bioresorbable afamelanotide implant from the optimized final manufacturing process.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Afamelanotide Group 1 (Experimental): A 16 mg bioresorbable afamelanotide implant (Group 1) from the previous manufacturing process.
  Interventions: Drug: Afamelanotide Group 1
- Afamelanotide Group 2 (Experimental): A 16 mg bioresorbable afamelanotide implant (Group 2) from the optimized final manufacturing process.
  Interventions: Drug: Afamelanotide Group 2

INTERVENTIONS:
Drug: Afamelanotide Group 1 — One 16 mg bioresorbable afamelanotide implant (Group 1) from the previous manufacturing process.
  Other Names: afamelanotide
  Arms: Afamelanotide Group 1
Drug: Afamelanotide Group 2 — One 16 mg bioresorbable afamelanotide implant (Group 2) from the optimized final manufacturing process.
  Other Names: afamelanotide
  Arms: Afamelanotide Group 2

SUMMARY:
This is a single center, pharmacokinetic and pharmacodynamic study in healthy volunteers. Twenty four subjects will be enrolled in the study and will be assigned to receive either a 16 mg afamelanotide bioresorbable implant from the current manufacturing process or a 16 mg afamelanotide bioresorbable implant from the optimized manufacturing process. Implants will be administered subcutaneously.

The following procedures will be conducted throughout the study:

* Collection of blood samples for analysis of afamelanotide concentrations
* Measurement of skin reflectance for estimation of melanin density, and luminance (L*), blue/yellow colour hue (b*)
* Safety monitoring

DETAILED DESCRIPTION:
The objective of the proposed study is to confirm that the pharmacokinetic and pharmacodynamic properties of implants eluting 16 mg of afamelanotide produced by this final optimized manufacturing process are essentially the same as those of implants manufactured with the same formulation that have been used in earlier clinical studies

The study will involve the use of an implant, which comes in the form of a small rod to be administered under the skin.

For this study, afamelanotide has been formulated as a controlled release depot injection (implant). This means that the afamelanotide will be released slowly into the body over a few days. Once inserted, the implant will remain in the body after afamelanotide has been released and will slowly dissolve.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Caucasian adults aged between 18 and 45 years (inclusive).
* Free of significant abnormal findings as determined during the screening procedure by surgical and medical history, physical examination, ECG, clinical laboratory testing and vital signs.
* BMI between 18 and 30 kg/m2 (inclusive).
* No history of drug abuse, licit or illicit (including alcohol).
* Agree not to use any medications (prescribed medicines, over-the-counter medications, dietary supplements or nutraceuticals) without pre-approval by the Principal Investigator or nominee during the 7 days preceding the study, and during the course of the study (until Day 60)
* Willing to take precautions to prevent pregnancy until completion of the study (Day 60).
* Able to understand and sign the written Informed Consent Form.
* Able and willing to follow the Protocol requirements, including refraining from the use of melanogenic (tanning) products and recreational sun or UV light exposure from the start of the study until Day 60

Exclusion Criteria:

* Any significant history of allergy and/or sensitivity to any of the contents of study drug product.
* Any significant history of allergy and/or sensitivity to lignocaine or other local anaesthetic.
* Any evidence of organ dysfunction or any clinically significant deviation from normal in the physical or clinical determinations.
* Personal history of melanoma, dysplastic nevus syndrome or family history of melanoma in a first degree relative.
* Any evidence at the screening medical examination of hypertension or hypotension. Hypertension is defined as three separate readings that persistently read over 140/90 mmHg systolic/diastolic. Hypotension is defined as three separate readings that persistently read under 90/50 mmHg systolic/diastolic.
* A pulse rate of less than 50 beats/minute.
* Any significant illness during the 4 weeks before the study screening period.
* Any contraindication to blood sampling.
* Any factor that may interfere with the skin reflectance measurements (e.g. vitiligo, albinism, excessive number of moles, or excessively hairy skin).
* Positive screening urine drugs of abuse test.
* Participation in any clinical study during the 4 weeks before the study screening period.
* Has donated 400 mL or more of blood or had significant blood loss during the 8 weeks preceding screening.
* Has donated plasma within the 7 days preceding screening.
* Have consumed alcohol during the 24 hours prior to Day 1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Change in skin melanin density | 120 days
  To confirm serial changes in skin melanin density by reflectance spectrophotometry following administration of the final formulation afamelanotide bioresorbable implants in healthy volunteers.

SECONDARY OUTCOMES:
Change in plasma concentrations of afamelanotide | 60 days
  To confirm the pharmacokinetics of afamelanotide by assessing afamelanotide plasma concentration following administration of the final formulation afamelanotide bioresorbable implants in healthy volunteers.
Number of Adverse Events | 60 days
  To confirm the tolerance of afamelanotide by assessing adverse events following administration of the final formulation afamelanotide implants in healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Matson, MD, Principal Investigator — Prism Research Inc.
Locations (1):
- Prism Research Inc., Saint Paul, Minnesota, United States